CLINICAL TRIAL: NCT02056509
Title: The Effect of Chest Compression and Ventilation Coordination During Cardiopulmonary Resuscitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201305100RINB
Record Dates: First submitted 2014-01-21; First posted 2014-02-06 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Out-of-Hospital Cardiac Arrest; Sudden Cardiac Death
Keywords: cardiopulmonary resuscitation,Ventilation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Death, Sudden, Cardiac; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Out of hospital cardiac arrest: Out of hospital cardiac arrest of non-traumatic cause
- Unexpected in-hospital cardiac arrest: Unexpected cardiac arrest during emergency department stay

SUMMARY:
Airway management and maintaining adequate ventilation during cardiopulmonary resuscitation (CPR) are important. The rule of 30:2 compression-to-ventilation ratios before endotracheal intubation and keeping 1 breath every 6-8 seconds with advanced airway are generally accepted according to 2010 Advanced Cardiac Life Support (ACLS) guideline. This recommendation emphasizes on the timing and frequency of ventilation during CPR. However, poor clinical evidence had been established concerning adequate volume, airway flow and pressure in each cycle.

There are increasing evidence that hyperventilation during resuscitation reduces pulmonary venous return and, therefore, compromises cardiac output and circulation. Another research reported that using high flow oxygen mask alone during basic life support (BLS) results in better survival rate and overall outcome compared with conventional positive pressure ventilation.

Our study applies flowmeter to measure ventilation parameters as frequency, duration, exhaled volume and airway pressure on intubated patients who received artificial ventilation during CPR. The parameters will correlate with information from accelerometry and capnometry simultaneously during resuscitation. . Investigators also focus on the influence of chest compression, which increases intra-thoracic pressure considerably. This effect may act against positive pressure ventilation and probably minimize the efficiency in each ventilation or circulation..

Details about how to ventilate one patient during CPR include right timing, duration, adequate volume and coordination are in debate. Unfortunately, current practice based on clinical guidelines emphasizes little on this issue. Investigators are committed to refine contemporary practices and hopefully improve qualities of resuscitation.

Investigators proposed the hypothesis that coordinate chest compression and ventilation may minimize the increasement of airway pressure and improve the effect of circulation

ELIGIBILITY:
Inclusion Criteria:

* age > 20 years old, < 100 years old

Exclusion Criteria:

* Trauma related out of hospital cardiac arrest

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiac arrest patient received CPR in Emergency Department Age > 20 years old
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
rate of 2- hour recover of spontaneous circulation | 2 hours
  Recover of spontaneous circulation lasting for 2 hours describe as successful recover of spontaneous circulation, otherwise failure.

SECONDARY OUTCOMES:
End tidal carbon-dioxide level | Measured during and end of resuscitation
  End tidal carbon-dioxide level correlates with successful recovery of spontaneous circulation event
Arterial blood gas data | measured during and end of resuscitaiton
  Oxygen and carbon-dioxide tension changes in different ventilation strategy in cardiopulmonary resuscitation
30-day survival rate | 30 days
90-day neurologic outcome | 90 days
Survive to discharge | 90 days
  Duration of hospital stay, usually will be recorded in 90 days, occasionally will more than 90 days
Timing of first shockable rhythm | measured during resuscitaion

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Chih Wang, Principal Investigator — Emergency department, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan